CLINICAL TRIAL: NCT00528593
Title: A Randomized, Multi-center Pilot Study to Evaluate the Efficacy and Safety of Epoetin Alfa (Procrit) in the Treatment of HIV-associated Sensory Neuropathy
Brief Title: Epoetin Alfa for HIV-Associated Neuropathy Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of pharmaceutical support
Sponsor: Washington University School of Medicine (Other)
Collaborators: Ortho Biotech Clinical Affairs, L.L.C. (Industry); PPD Development, LP (Industry); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: David B. Clifford, M.D., Principal Investigator, Neurologic AIDS Research Consortium, Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U01 NS32228- ninds; U01NS032228 (NIH)
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: HIV Infections; Neuropathy
Keywords: HIV; AIDS; neuropathy; Procrit; epoetin alfa; erythropoetin; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Epoetin Alfa; Erythropoietin

ARMS (1):
- 1 (Active Comparator)
  Interventions: Drug: epoetin alfa

INTERVENTIONS:
Drug: epoetin alfa — Group 1 will receive Procrit once every three weeks, and group 2 will receive Procrit every week.
  Other Names: Procrit; erythropoetin

SUMMARY:
The purpose of this study is to evaluate the effect of epoetin alfa on HIV-associated neuropathy by measuring changes in nerve fiber density and pain ratings.

DETAILED DESCRIPTION:
The Neurologic AIDS Research Consortium (NARC) designs and carries out clinical trials to improve the therapy for HIV induced neurologic disease, and neurologic conditions associated with the AIDS virus.

Complications of HIV are dynamically evolving over time. In general, neurologic complications that typically occur in advanced disease stages are increasing in incidence while some of the early complications associated with AIDS are less commonly found due to improved preventive therapy. The impact of the new generation of antiretroviral drugs, and of predominantly multi-drug therapy remain to be seen. Several key new drugs fail to penetrate the brain, thus making it possible for the incidence of neurologic disease to continue to increase. NARC develops studies based on the current challenges of the AIDS epidemic.

Erythropoetin (also known as epoetin alfa or Procrit) is naturally produced in the body. Procrit or epoetin alfa is an injectable form of synthetic erythropoietin. In this trial, scientists will evaluate the effect of epoetin alfa on HIV-associated neuropathy by measuring changes in nerve fiber density and pain ratings. The goal of the trial is to determine if epoetin alfa increases the number of nerve fibers in the skin of people with HIV-associated neuropathy, and improves symptoms of neuropathy. This study will also find out if Procrit is safe and well-tolerated for treating the painful neuropathy associated with HIV.

After two screening visits, participants will be randomly assigned to one of two groups: group 1 will receive Procrit once every three weeks, and group 2 will receive Procrit every week. Follow-up treatment visits will occur at weeks 6, 12, 24, 36, and 48. During the visits, participants will have their blood pressure and heart rate measured. During several of the follow-up visits participants will be asked to rate the intensity of their pain using the Gracely Pain Scale and the McGill Pain Questionnaire. Duration of this trial for participants is 52 weeks or 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or female ≥ 18 years old.
* Subject has documented HIV-1 infection.
* Subject has stable use or no use of specific dideoxynucleoside reverse transcriptase inhibitors (ie. ddI, d4T, ddc) for ≥4 months prior to Visit 1.
* Subject has painful HIV-associated sensory neuropathy (either DSP or ATN), as confirmed by a neurologist.
* Subject has an average severity of neuropathic pain over the 2 week period between visit 2 and Visit 3 of ≥0.74 units measured with the Gracely pain intensity scale.
* Subject (either male or female) agrees not to participate in a conception process (i.e. active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization), and use of contraception.
* Subjects hemoglobin is less than 13.0g/dl but greater than or equal to 10.0g/dl.

Exclusion Criteria:

* Subject has any condition other than HIV infection or antiretroviral therapy that in the opinion of the site neurologist confounds the diagnosis of neuropathy.
* Subject has received insulin or oral hypoglycemic products for treatment of diabetes mellitus £30 days from Visit 1.
* Subject has a documented history of untreated vitamin B12 deficiency (serum B12 level less than 200 pg/mL) or less than 3 months of B12 supplementation (injection or intranasal B12) prior to screening. Use of a multivitamin is permissible.
* Subject has hereditary neuropathy or compression-related neuropathies, i.e. spinal stenosis, that would preclude analysis of treatment response.
* Subject has received treatment with any drug other than the dideoxynucleoside analogues that the site neurologist considers to have significantly contributed to the subject's neuropathy ≤30 days from Visit 1.
* Subject has a history of any alcohol-related medical complications within 6 months of Visit 1 including, but not limited to, alcohol withdrawal seizures, hallucinosis, delirium tremens, or being in a detoxification program.
* Subject has received neurotoxic chemotherapeutic agents £90 days from Visit 1.
* Subject has received neuroregenerative agents £90 days from Visit 1.
* Subject has myelopathy that would interfere with the evaluation of the subject.
* Subject has uncontrolled hypertension (Systolic Bp>160mmHg and/or Diastolic Bp >100mmHg)
* Subject has known hypersensitivity to mammalian cell-derived products or albumin.
* Subject has a history of thrombotic events or epileptic seizures.
* Subject has an active AIDS-defining opportunistic infection (OI) or OI-defining condition £30 days from Visit 1.
* Subject has active major disease, both HIV-related and non-HIV-related including, but not limited to, cardiac disease, pulmonary, or hepatorenal, which in the opinion of the investigator might affect the study.
* Subject is pregnant or breast-feeding.
* Subject has any currently active malignancy, or a history of any previous malignancy with the exception of skin squamous cell carcinoma or basal cell carcinoma.
* Subject has received any investigational agent(s) that is not FDA-approved or has participated in any interventional research study £30 days from Visit 1.
* Subject is actively using recreational intravenous drugs, crack cocaine, or intranasal/smoked heroin or methamphetamine.
* Subject has chronic renal failure defined for the purposes of this study as a creatinine >1.5 x upper limit of normal (ULN).
* Subject has hepatitis C and is on interferon/ribavirin therapy or interferon/ribavirin therapy is planned over the expected course of the study.
* Subject has received epoetin alfa (Procrit) within 2 months prior to study entry.
* Subject has HgbA1C >6.5.
* Subject has serum B12 ≤200 pg/mL.
* Subject has hemoglobin <11.0 g/dL.
* Subject has INR >1.4 or platelets <50,000.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Difference between the distal leg intra-epidermal nerve fiber density | at baseline and after 48 weeks of treatment

SECONDARY OUTCOMES:
Change in pain levels measured via Gracely pain scale between baseline and every 6 weeks thereafter up to 48 weeks | up to 48 weeks
Change in global physician impression from the Visit 4 baseline measurement and measurement after 48 weeks of treatment | baseline and after 48 weeks of treatment
Differences between Quantitative Sensory Testing measurement at baseline and after 48 weeks of treatment | at baseline and after 48 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Justin McArthur, MBBS, MPH, Study Chair — Professor of Neurology, Johns Hopkins University; David B. Clifford, MD, Principal Investigator — Professor of Neurology, Washington University; David Simpson, MD, Principal Investigator — Professor of Neurology, Mt. Sinai Medical Center; Bruce Cohen, MD, Principal Investigator — Professor of Neurology, Northwestern University; Pablo Tebas, MD, Principal Investigator — Associate Professor of Medicine, University of Pennsylvania